CLINICAL TRIAL: NCT02587780
Title: An Observational Study of Incremental Area Under the Curve Values in Similar, Non-diabetic, Subjects- Undertaking Different Amounts and Intensities of Physical Activity
Brief Title: Blood Sugar Responses by Physical Activity Level and Intensity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Small Changes (Other)
Collaborators: Sheffield Hallam University (Other)
Responsible Party: Sponsor
Other Study IDs: SBSREC1314/37
Record Dates: First submitted 2015-10-02; First posted 2015-10-27 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Inactive: people who perform < 30mins.day physical activity at a 'moderate' level of intensity.
- Active: people who perform 30mins-60 mins.day of physical activity at a 'moderate' level of intensity.
- Very active: People who perform > 60 mins.day of physical activity at a >moderate level of intensity.

SUMMARY:
This observational study is designed to examine the glycaemic responses (of sedentary, active and very active healthy individuals) to a 50gram dose of glucose.

DETAILED DESCRIPTION:
3 groups of participants fulfilling the criteria for: sedentary (< 30mins phys activity p/day) active (>30 mins phys act p/day) and very active (> 60 mins phys act p.day) will be invited to attend a laboratory session on two separate occasions separated by one week and asked to: fast overnight before having a baseline and then six further capillary (finger-prick) blood samples taken over a period of two hours following consumption of 50 grams of glucose. The blood samples will produce a standard glucose 'curve' and this will be used to calculate incremental area under the curve to identify similarities or differences between the three groups responses. Hypothetically it may be that the different levels and intensities of physical activity will affect the results with active individuals producing flatter better-controlled blood sugar responses than the inactive subjects. The Null-hypothesis would be no difference in response. it is possible, for instance, that such a low-dose of glucose in an otherwise healthy group of individuals has no discernible affect on such a curve. Physical activity will be assessed by questionnaire and interview. Anthropometric measures (height, weight and body composition) will be taken using a stadiometer and bio-electrical impedance unit (Bodystat 1500, Body Stat: Isle of man UK) at the time of the laboratory measures. No participants will have data taken of any kind before they have read a participant information sheet and signed informed consent.

ELIGIBILITY:
Inclusion Criteria:

* male and female.
* age:19-59
* inactive, active or very active according to criteria outlined.

Exclusion Criteria:

* Diabetics other chronic condition likely to affect blood sugar
* <19>59 age

Ages: 19 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy individuals (non-diabetic or other chronic disabling conditions likely to affect blood glucose) of different habitual levels of physical activity.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2015-11; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Blood glucose response | One year
  blood glucose responses in sedentary, active and very active groups of men and women

SECONDARY OUTCOMES:
Body mass index | One year
  Height in metres squared divided by weight in kilograms
Physical Activity duration | One year
  A questionnaire to asses daily physical activity participation
Intensity of physical activity | One year
  A questionnaire assessing rating of perceived exertion
Body fat percentage | One year
  percentage body fat recorded by bio-electrical impedance